CLINICAL TRIAL: NCT06273462
Title: Randomized Placebo-Controlled Trial of Palmitoylethanolamide for Chronic Inflammatory Pain Conditions
Brief Title: Palmitoylethanolamide for Chronic Inflammatory Pain Conditions
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Navy Medical Center San Diego (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NMCSD.2024.0006
Record Dates: First submitted 2024-02-06; First posted 2024-02-22 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Chronic Pain
Keywords: chronic pain; supplement; alternative therapy
MeSH Terms: conditions — Chronic Pain | interventions — palmidrol

STUDY DESIGN:
Intervention Model Description: Prospective Randomize Double Blind Placebo Controlled study comparing the supplement palmitoylethanolamide (PEA) to a visually identical placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blinded, patients will receive visually identical capsules from research pharmacist with study label indicating PEA vs Placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Palmitoylethanolamide (Experimental): Participants randomized to the experimental arm will receive the supplement Palmitoylethanolamide (PEA) at a dose of 600mg twice a day
  Interventions: Drug: Palmitoylethanolamide 600mg twice a day
- Placebo (Placebo Comparator): Participants randomized to the placebo arm will receive a visually identical placebo capsule
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Palmitoylethanolamide 600mg twice a day — 600mg palmitoylethanolamide twice a day
  Other Names: PEA
  Arms: Palmitoylethanolamide
Other: placebo — visually identical placebo capsule
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate if a supplement called palmitoylethanolamide (PEA) is effective in reducing the pain in patients with chronic inflammatory pain conditions. The main question the trial aims to answer is if PEA works better at treating a patients pain and improving their function better than a placebo.

Participants will be divided into two equal groups and asked to take either PEA or a placebo for 8 weeks.

DETAILED DESCRIPTION:
Chronic inflammatory pain conditions, such as rheumatoid arthritis, fibromyalgia, and neuropathic pain syndromes, present a significant burden on individuals and healthcare systems worldwide. Despite advancements in pain management, many patients continue to experience inadequate relief, and the long-term use of conventional analgesics can be associated with adverse effects.

Palmitoylethanolamide (PEA) is a naturally occurring fatty acid amide that has garnered attention in recent years for its potential therapeutic properties in managing chronic inflammatory pain. PEA is an endogenous lipid mediator and a member of the N-acylethanolamine family. It exerts its effects primarily by interacting with peroxisome proliferator-activated receptor alpha (PPAR-α) and through other molecular pathways involved in neuroinflammation and immune responses.

In Europe where nutraceuticals are more commonly used in conventional practice, research on PEA has shown significant promise in studies on inflammatory pain conditions such as chronic pelvic pain, irritable bowel syndrome, temporomandibular joint arthritis and knee osteoarthritis. Similar studies have not been completed in the United States.

1. Anti-Inflammatory Effects:

   - PEA has demonstrated anti-inflammatory properties by modulating immune responses, inhibiting mast cell activation, and reducing the release of pro-inflammatory cytokines. These effects suggest its potential in attenuating the underlying inflammation in chronic pain conditions.
2. Analgesic Effects:

   - Several animal studies have reported that PEA can alleviate pain in models of neuropathic pain, inflammatory pain, and even in more complex pain conditions like fibromyalgia. These findings suggest that PEA may have a role as an analgesic agent.
3. Safety and Tolerability:

   - PEA is generally well-tolerated with a favorable safety profile. Clinical trials and real-world studies have reported minimal side effects, making it a potentially attractive option for long-term use in chronic pain management.
4. Clinical Trials:

   - Some clinical trials have explored the use of PEA in specific chronic pain conditions. While results have been promising, larger, well-controlled trials are needed to establish its efficacy conclusively.
5. Mechanisms of Action:

   * Beyond PPAR-α activation, PEA may also influence other cellular pathways involved in pain modulation, such as TRPV1 channels and GPR55 receptors, although the exact mechanisms are still being elucidated.

Summary of previous trials:

A recent systematic review and meta-analysis of no US studies suggests that PEA is an effective and well-tolerated treatment for chronic pain. The literature search identified 253 unique articles with 11 included in the meta-analysis. The 11 articles had a combined sample size of 774 patients with diverse chronic pain conditions who took a dose of 400-1200 mg of a PEA supplement or a placebo over periods ranging from 2 to 12 weeks. The studies showed significantly better pain reduction compared to placebo with no adverse effects.

Given the growing interest in PEA as a potential therapeutic agent for chronic inflammatory pain, and the lack of any known side effects of this supplement, this randomized placebo-controlled trial aims to contribute valuable data to the existing body of research. By rigorously evaluating the efficacy and safety of PEA in a controlled clinical setting, the investigators seek to provide evidence-based insights into its role in managing chronic inflammatory pain conditions and further inform clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Inflammatory Pain of greater than 3 months duration and greater than or equal to 5/10 intensity that has not responded to other conservative therapies such as rest, ice, compression or other oral medications.

Exclusion Criteria:

* Severe allergy to any specific food component such as nut, egg or soy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-08-05 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Pain Level | 4 and 8 weeks
  Pain level will be assessed using the Defense and Veterans Pain Rating Scale (DVPRS) Where the minimum value is 0 indicating no pain and the maximum value is 10 indicating worst possible pain

SECONDARY OUTCOMES:
Pain interference and function | 4 and 8 weeks
  Daily Pain Impact (interference with activity, sleep, mood, stress) (0-10 scale with 0 being the best and 10 being the worst outcome)
Pain Catastrophizing Scale (PCS) | 4 and 8 weeks
  Pain Catastrophizing Scale (PCS) (Helplessness; Magnification; Rumination) (0-52 scale with 0 being the best and 52 being the worst outcome)
Patient Reported Outcome Measurement Information System (PROMIS) (Pain interference, Social satisfaction; Physical function) | 4 and 8 Weeks
  PROMIS (Pain interference, Social satisfaction; Physical function) (0-10 each with 0 being the worst and 10 being the best outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States